CLINICAL TRIAL: NCT04588909
Title: Outcomes of Elective Colorectal Cancer Surgery During COVID 19 Pandemic: Implications for Cancer Care Policy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheri Kashmir Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, ASIF MEHRAJ, Senior Resident, Sheri Kashmir Institute of Medical Sciences
Other Study IDs: 73/2020 (Supl 2)
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Colo-rectal Cancer
Keywords: colorectal cancer; COVID 19 pandemic
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colorectal resections — All patients admitted with colorectal cancer were subjected to various types of colorectal resections

SUMMARY:
Due to COVID 19 (Corona virus disease)pandemic, majority of surgeries, including surgery for cancer patients got delayed across the globe. Surgeries were limited to emergency set up only. At our institute we tried to perform colorectal cancer surgeries through out the pandemic, albeit in less numbers, as we thought cancer in itself is an emergency setting. we are planning to analyse the prospectively managed database of this particular group of patients over a period of last six 6 months and look out at 30 day post operative morbidity and mortality. Besides we will try to analyse the implications of our decision to carry on with cancer surgeries in terms of number of health care workers who got infected while being involved in primary care of these patients.

DETAILED DESCRIPTION:
INTRODUCTION Health systems all across the globe have been under tremendous stress due to COVID 19 pandemic. Based on information suggesting that India was faring better compared to the west [1] and that oncology patients were likely to get deferred care with significant implications [2], the department of general surgery (colorectal division) took a conscious decision to continue offering elective cancer surgeries albeit in less numbers.in this study we will try to collect 30 day post operative outcome data of elective colorectal cancer resections at our department and discuss the implications of our decision.

Such reports are still sparsely reported from Covid hotspots around the world.

Methods:

We will analyze the prospective database of the department of colorectal surgery at Sheri Kashmir Institute of Medical Sciences, Srinagar, a tertiary referral centre and a high volume centre for colorectal cancer surgeries ( with more than 300 colorectal cancer surgeries performed every year) in North India wef 23rd March to 22nd September 2020 (6 months).and report outcomes of all elective colorectal cancer surgeries. Each patient will be followed up for 30 days, thereby last follow up will end on 22nd October 2020.

All colorectal cancer patients subjected to elective and emergency surgeries during COVID 19 pandemic will be included. Patients who were positive for SARS CoV2 (Severe acute respiratory syndrome coronavirus 2) infection and underwent surgery for colorectal cancer will be excluded.

The data will be statistically analysed using Statistical Product and Statistical Solutions(SPSS) sotware v 23. All categorical variables will be shown in the form of frequency and percentage. Continuous variables will further be analysed by independent t test and using multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer patients subjected to surgery during COVID 19 pandemic

Exclusion Criteria:

* SARS CoV 2 infected patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Colorectal cancer patients subjected to both elective and emergency surgery during COVID 19 pandemic.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-10-22 (Estimated)

PRIMARY OUTCOMES:
Early post operative mortality | 30 days
  patients who died within 30 days following their surgery

SECONDARY OUTCOMES:
Early Post operative complications | 30 days
  post operative complications will be graded as per clavien dindo grading system
Incidence of SARS CoV2 infectivity among health care providers providing direct care to involved patients | 30 days
  determine whether any health care worker involved with the care of this cohort of patients got infected with SARS CoV 2.
Rate of hospital acquired SARS CoV 2 infection among operated patients. | 30 days
  Determine whether any patient from the cohort got infected with SARS CoV 2 during their hospital stay or immediately after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nisar A Chowdri, Study Chair — Government organisation
Locations (1):
- Sher i Kashmir Institute of Medical Sciences, Srinagar, Jammu and Kashmir, India

IPD SHARING:
Plan to Share IPD: No